CLINICAL TRIAL: NCT06995495
Title: Wearable Device for Characterizing AMI Patients After Primary PCI and Predicting the Clinical Outcomes
Brief Title: Wearable Devices Faciliate the Management of AMI Patients
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhiguo Zou, Doctor, RenJi Hospital
Other Study IDs: EARLY-MYO Wearable Devices
Record Dates: First submitted 2025-01-21; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will explore the use of wearable technology to consistently monitor patients with acute myocardial infarction (AMI) receiving primary percutaneous coronary intervention (PCI). Parameters such as heart rate, sleep time, physical activity, and blood pressure will be collected and analyzed to characterize the patients and predict clinical outcomes.

DETAILED DESCRIPTION:
The aim of this study is to explore in-hospital patient management and predict clinical outcomes in AMI patients receiving primary PCI through wearable technology (e.g., smart watches and wristband devices). The investigators expect to involve patients diagnosed with AMI, including ST-elevation myocardial infarction (STEMI) and non-ST-elevation myocardial infarction (NSTEMI), who are admitted to the cardiac Cardiac Intensive Care Unit (CICU) after primary PCI.

With written consent, eligible participants will be consistently monitored by a wearable device during the CICU stay, in addition to a conventional monitoring system. Vital signs including heart rate (beats/minute), oxygen saturation (%) blood pressure (mmHg), and other crucial parameters such as sleep patterns will be recorded. The collected data will be analyzed using AI-assisted and machine learning techniques, integrated with other clinical data to construct models that support risk stratification, guide clinical decision-making, improve the quality of nursing care, and predict long-term prognosis for these patients. Serial follow-ups (6-month, annual, and long-term) will be performed, and important information such as cardiac function assessed by echocardiography, the incidence of major adverse cardiovascular events, and life qualities will be collected for each follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old
* Diagnosed with STEMI or NSTEMI (ACC/AHA guidelines)
* Half male and half female
* Undergo CAG and PCI treatment;
* Written informed consent.

Exclusion Criteria:

* People under the age of 18 years old;
* Patients who are pregnant/breastfeeding;
* Patients who are allergic to the metallic or plastic components of the wearable devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with AMI, including ST-elevation myocardial infarction (STEMI) or non-ST-elevation myocardial infarction (NSTEMI), and admitted to cardiac Cardiac Intensive Care Unit (CICU) after primary PCI.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Pattern assessed artificial intelligence (AI)-assisted analysis | Throughout the full course of hospitalization, with an average of 1 week.
  The dynamic trajectory or trend of a patient's heart rate measurements over the course of hospital stay. Time series data will be analyzed by AI-assisted machine learning model.

SECONDARY OUTCOMES:
Cardiac function assessed by echocardiography | At 1-month, 6-month and 1-year follow-ups.
  Cadiac function is evaluated as left ventricular ejection fraction (LVEF, %) by echocardiography
The event rate of coronary revascularization | From date of enrollment until the date of follow-ups at 1-month, 6-month and 1-year post discharge.
  The proportion (%) of participants who undergo an unplanned coronary revascularization procedure-either percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
The event rate of heart failure | From date of enrollment until the date of follow-ups at 1-month, 6-month and 1-year post discharge.
  The proportion (%) of participants who experience symptomatic heart failure. Heart failure is diagnosed based on symptoms such as shortness of breath and excess fluid, in the presence of a reduced LVEF (<60%) as assessed by echocardiography.
The event rate of re-infarction | From date of enrollment until the date of follow-ups at 1-month, 6-month and 1-year post discharge.
  The proportion (%) of participants who experience recurrent myocardial infarction, refers to a new or additional heart attack that occurs after the myocardial infarction diagnosed at enrollment.
Cardiovascular mortality (%) | From date of enrollment until date of death from cardiovascular causes, or assessed up to 12 months.
  Cardiovascular mortality (%) is defined as the proportion of participants who die due to cardiovascular causes during the follow-up period. Cardiovascular causes include myocardial infarction, heart failure, stroke, sudden cardiac death, or other documented cardiac or vascular events.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China